CLINICAL TRIAL: NCT03593395
Title: LCI-HEM-SCD-ST3P-UP-001: A Comparative Effectiveness Study of Peer Mentoring [PM] Versus Structured Transition Education Based Intervention [STE] for the Management of Care Transitions in Emerging Adults With Sickle Cell Disease (SCD)
Brief Title: LCI-HEM-SCD-ST3P-UP-001: The Sickle Cell Trevor Thompson Transition Project (ST3P-UP Study)
Acronym: ST3P-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: LCI-HEM-SCD-ST3P-UP-001; 00027706 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2018-06-14; First posted 2018-07-20 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: Sickle Cell Disease
Keywords: Transition; Emerging Adults; Peer Mentoring
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Parallel group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program Structured Education Based Transition Program (Active Comparator): Program Structured Education Based Transition Program [STE]
  Interventions: Other: Structured Education Based Transition Program STE
- Structured Education Based Transition Program + Peer Mentoring (Experimental): Structured Education Based Transition Program [STE] + Peer Mentoring [PM]
  Interventions: Other: Peer Mentoring [PM]; Other: Structured Education Based Transition Program STE

INTERVENTIONS:
Other: Peer Mentoring [PM] — Virtual Peer Mentoring
  Arms: Structured Education Based Transition Program + Peer Mentoring
Other: Structured Education Based Transition Program STE — Education-based program

SUMMARY:
This multi-center study will compare the effectiveness of adding virtual peer mentoring (PM) to a structured education-based (STE) transition program for emerging adults with sickle cell disease to determine its effect on decreasing the number of acute care visits per year, improving patient-reported outcomes, and reducing healthcare utilization among emerging adults with sickle cell disease (EA-SCD)

DETAILED DESCRIPTION:
This is a multi-center, cluster randomized study comparing the effectiveness of adding virtual peer mentoring (PM) to a structured education-based (STE) transition program based on the 6 core elements of transition in improving acute care reliance, quality of life and satisfaction with transition process in emerging adults with sickle cell disease (EA-SCD). The study will involve a total of 14 large (>80 EA-SCD currently in pediatric care) and small-scale (≤80 EA-SCD currently in pediatric care) clinical sites, with a 1:1 randomization at the site level. The study will involve approximately 700 subjects, 120 peer mentors, and 25 advisors. The primary endpoint of this study will be the average number of acute care visits per year over a minimum of 24 months. Secondary objectives are to compare the effectiveness of STE+PM versus STE alone at improving patient-reported outcomes and reducing healthcare utilization among EA-SCD. Enrollment is anticipated to occur over 18-24 months

ELIGIBILITY:
EA-SCD Eligibility Criteria:

Inclusion Criteria:

* Age 16 and < 25 years at the time of consent AND being cared for in a PEDIATRIC SICKLE CELL PROGRAM
* Any sickle cell genotype
* Not known to be currently pregnant
* Ability to read and understand the English language
* Subject is planned to be transferred to an adult sickle cell program within 6-12 months of consent

Exclusion Criteria:

* Already receiving one on one peer mentoring as part of a transition program -As determined by the Investigator, uncontrolled undercurrent medical, psychiatric, or cognitive condition, or social situation that would limit compliance with study requirements
* Pregnant, incarcerated, or otherwise unable to attend all study related visits
* Lack of easy access to the technology required to complete study surveys (e.g., internet in home setting, public area or at local CBO) or to conduct mentoring sessions
* Other factors that would cause harm or increase risk to the participant or close contacts, or preclude the participants adherence with or completion of the study.

Mentor Eligibility Criteria:

* Be an adult living with SCD or a caregiver of an adult living with SCD who has successfully transitioned to adult care (defined as having had at least 3 visits or a year of continuous care with an adult sickle cell provider)
* Age 26-35 years
* Readily available access to a computer with internet
* Have completed and passed a background check
* Legally able to work in the United States
* Ability to read and understand the English language
* Endorsed by their healthcare provider as reliable and able to meet the physical, psychological and cognitive requirements for serving as a mentor

Advisor Eligibility Criteria:

* Be an adult living with SCD or a caregiver of an adult living with SCD who has successfully transitioned to adult care (defined as having had at least 3 visits or a year of continuous care with an adult sickle cell provider)
* Age ≥ 36 years
* Readily available access to a computer with internet
* Have completed and passed a background check
* Ability to read and understand the English language
* Endorsed by their healthcare provider as reliable and able to meet the physical, psychological and cognitive requirements for serving as an advisor

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Payal Desai, MD, Principal Investigator — Wake Forest University Health Sciences; Raymona Lawrence, DRPH, Principal Investigator — Wake Forest University Health Sciences
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Health System, Mobile, Alabama
  - University of Miami, Miami, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Greenville Health System, Greenville, South Carolina
  - Virginia Commonwealth University (VCU), Richmond, Virginia

REFERENCES:
- [Background] Osunkwo I, Lawrence R, Robinson M, Patterson C, Symanowski J, Minniti C, Bryant P, Williams J, Eckman J, Desai P. Sickle Cell Trevor Thompson Transition Project (ST3P-UP) protocol for managing care transitions: Methods and rationale. Contemp Clin Trials. 2023 Mar;126:107089. doi: 10.1016/j.cct.2023.107089. Epub 2023 Jan 18. PMID 36669729

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Site
Period: Overall Study
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Started | 196; 7 Site | 95; 7 Site
Completed | 121; 7 Site | 49; 7 Site
Not Completed | 75; 0 Site | 46; 0 Site
Not completed — Lost to Follow-up | 48 | 3
Not completed — Withdrawal by Subject | 5 | 24
Not completed — Death | 2 | 3
Not completed — Physician Decision | 0 | 6
Not completed — Participant Relocated | 19 | 3
Not completed — No Information | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring | Total
Number analyzed (Participants) | 196 | 95 | 291
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.9 (1.4) | 18.7 (1.7) | 18.8 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 51 | 151
  Male | 96 | 44 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 182 | 90 | 272
  Unknown or Not Reported | 6 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 188 | 90 | 278
  Race: Other | 6 | 5 | 11
  Race: Unknown | 2 | 0 | 2
Acute Care Visits per Year (Historical) [Mean (Standard Deviation); unit: visits per year] | 4.0 (5.2) | 2.6 (4.3) | 3.6 (4.9)
Ambulatory Care Visits per Year (Historical) [Mean (Standard Deviation); unit: visits per year] | 5.9 (7.3) | 7.0 (5.5) | 6.3 (6.8)
SCD Phenotype [Count of Participants; unit: Participants]
  SS Disease | 134 | 60 | 194
  SC Disease | 45 | 18 | 63
  Other | 17 | 17 | 34
Overall PedsQL SCD Score (0-100) [Mean (Standard Deviation); unit: units on a scale] — PedsQL SCD - Pediatric Quality of Life Sickle Cell Disease Module. Indicates patient's perception of their quality of life. Higher score is better. 43 items, 9 dimensions: Pain and Hurt, Pain Impact, Pain Management, Worry I, Worry II, Emotions, Treatment, Communication I, Communication II. Individual questions are scored on 5-point Likert scale, (0=never, 4=almost always); scores are transformed on a scale from 0-100, (0=100, 1=75, 2=50, 3=25, 4=0). If >50% of items are missing, scale scores are not computed. If >=50% items are completed, mean of completed items is imputed for total score. Population: Data presented for those who completed the survey.
  units on a scale
    number analyzed (Participants) | 150 | 59 | 209
    (all) | 63.2 (18.4) | 61.3 (19.6) | 62.6 (18.7)
Overall MOS-SSS Score (0-100%) [Mean (Standard Deviation); unit: units on a scale] — MOS-SSS - Medical Outcomes Study Social Support Survey. Patient's perceived social support score. Higher score indicates more support. 19 items, 4 subscales plus overall functional social support index. Each item is 5-level Likert scale (1=None of the time, 5=All of the time). For each of subscales, respondent-specific mean scores are calculated, ignoring items with missing values. If >=1 valid response is available on subscale, a score is computed for that subscale. To calculate overall total, take average of item scores for completed items and transform to a 0-100 scale. Population: Data presented for those who completed the survey
  units on a scale
    number analyzed (Participants) | 155 | 61 | 216
    (all) | 75.3 (22.8) | 70.7 (24.1) | 74.0 (23.2)
Overall TIP-RFT Score (0-88) [Mean (Standard Deviation); unit: units on a scale] — TIP-RFT - Transition Intervention Program Readiness for Transition. Indicates patient's readiness to transition. A lower score indicates higher readiness. TIP-RFT includes 22 items, 4 subscales (Independent Living Skills, Healthcare Knowledge and Skills, Education and Vocational Planning, Social Support Skills). For total TIP-RFT, use sum of scales, total score range (0-88), smaller score is better. If any items were missing, the scores were not computed. Population: Data presented for those who completed the survey.
  units on a scale
    number analyzed (Participants) | 120 | 55 | 175
    (all) | 14.8 (11.0) | 12.9 (9.6) | 14.2 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Acute Care Visits (Visits Per Year)
Description: Acute care visits was calculated for each patient as the number of acute care visits over the duration of follow-up (time from enrollment to discontinuation of study participation). Acute visits were identified by manual chart reviews and included hospital admissions, ED, urgent care, day hospital, or infusion center visits. Acute care visits were calculated as the total number of acute care visits reported on study over the years the subject was on study.
Time Frame: Duration of time on study, on average 23 months
Population: All enrolled subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: visits per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 196 | 95
visits per year | 2.46 [1.81 to 3.34] | 2.96 [2.09 to 4.19]
Statistical Analysis 1: Comparison: Program Structured Education Based Transition Program; Test type: Other — Estimation only; Least Square Mean Estimate = 2.46, 95% CI 2-sided [1.81 to 3.34] — Estimates are from generalized linear mixed model with a negative binomial distribution log link construct and length of follow up offset. Includes fixed effects for site size, baseline acute utilization, and random effect for cluster (site)
Statistical Analysis 2: Comparison: Structured Education Based Transition Program + Peer Mentoring; Test type: Other — Estimation only; Least Square Mean Estimate = 2.96, 95% CI 2-sided [2.09 to 4.19] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Overall Rating of Health Care From Adults Sickle Cell Quality of Life Measurement Information System Quality of Care Measure (ASCQ-ME QOC)
Description: Specific item from ASQC-ME QOC. The survey measures patients' self-reported levels of quality of care received. This item was scored on a 10-point scale categorized to three ranges (0-6, 7-8, and 9-10). A "0" value is least, and a "10" value is best. 0-6 indicate the worst care, 7-8 indicate average care, 9-10 indicate the best care. Higher score indicates higher quality of care.
Time Frame: 6 and 12 months post-enrollment.
Population: Among participants with survey data available at relevant time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 80 | 26
Participants
  6 months: number analyzed (Participants) | 80 | 25
  6 months: 0-6 | 4 | 4
  6 months: 7-8 | 26 | 5
  6 months: 9-10 | 50 | 16
  12 months: number analyzed (Participants) | 55 | 26
  12 months: 0-6 | 10 | 3
  12 months: 7-8 | 17 | 6
  12 months: 9-10 | 28 | 17

3. Secondary Outcome: Pediatric Quality of Life - Sickle Cell Module (PedsQL-SCD Module) for Health-related Quality of Life
Description: Overall patient's perception of their quality of life. Higher quality of life score is better. There are 43 items with 9 dimensions: Pain and Hurt, Pain Impact, Pain Management, Worry I, Worry II, Emotions, Treatment, Communication I, Communication II. Individual questions are scored on a 5-point Likert scale, (0=never, 4=almost always) and scores are transformed on a scale from 0-100, where 0=100, 1=75, 2=50, 3=25, 4=0. If more than 50% of the items are missing, the scale scores should not be computed. If 50% or more items are completed, the mean of the completed items is imputed for the total score.
Time Frame: At 6 and 12 months post-enrollment
Population: Participants with data at 6 and 12 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 82 | 27
score on a scale
  6 months: number analyzed (Participants) | 82 | 26
  6 months | 66.5 [63.5 to 69.4] | 63.4 [58.0 to 68.8]
  12 months: number analyzed (Participants) | 58 | 27
  12 months | 68.7 [65.3 to 72.1] | 62.4 [57.2 to 67.6]

4. Secondary Outcome: Medical Outcomes Study Social Support Survey (MOS-SSS) Overall Social Support
Description: Patient's perceived social support score. A higher score for an individual scale or for the overall support index indicates more support. MOS-SSS includes 19 items, with four separate social support subscales and an overall functional social support index. Each item is a 5-level Likert scale (1=None of the time, 5=All of the time). For each of the 4 subscales, respondent-specific mean scores are calculated, ignoring items with missing values. If at least one valid response is is available on a subscale, a score can be received for that subscale. To calculate overall total, take average of item scores for completed items and transform to 0-100 scale (100 is best possible outcome).
Time Frame: At 6 and 12 months post-enrollment.
Population: Participants who completed the survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 84 | 28
score on a scale
  6 Months: number analyzed (Participants) | 84 | 27
  6 Months | 76.8 [71.8 to 81.7] | 77.8 [70.1 to 85.5]
  12 Months: number analyzed (Participants) | 64 | 28
  12 Months | 75.3 [70.0 to 80.7] | 80.6 [73.2 to 88.0]

5. Secondary Outcome: Transition Intervention Program Readiness for Transition (TIP-RFT) Scale
Description: Patient's readiness to transition scale. A lower score indicates higher readiness. TIP-RFT includes 22 items, with 4 subscales: (1) Independent Living Skills (8 items, range 0-32), (2) Healthcare Knowledge and Skills scale (6 items, range 0-24), (3) Education and Vocational Planning scale (4 items, range 0-16), (4) Social Support Skill set (4 items, range 0-16). For total TIP-RFT, use sum of scales. Total score range (0-88), smaller score is better. If any items were missing, the scores were not computed.
Time Frame: At 6 and 12 months post-enrollment.
Population: Participants who completed the survey.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 80 | 28
score on a scale
  6 Months: number analyzed (Participants) | 80 | 27
  6 Months | 10.4 [8.3 to 12.5] | 8.5 [4.9 to 12.1]
  12 Months: number analyzed (Participants) | 62 | 28
  12 Months | 9.4 [7.0 to 11.7] | 8.0 [4.7 to 11.3]

6. Secondary Outcome: Health Care Transition Feedback Survey Item: How Often Does Your Health Care Provider Explain Things in a Way That is Easy to Understand?
Description: Specific item from the Health Care Transition Feedback Survey, created by Got Transition. The survey evaluated patients' experience with changing from a pediatric to an adult approach to care. This question evaluated how often the health care provider explained things in a way that was easy to understand. Answer categories for this item were Always, Usually, Sometimes, and Never.
Time Frame: 12 months post-enrollment.
Population: Participants with survey data at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 51 | 26
Participants
  Always/Usually | 48 | 26
  Sometimes/Never | 3 | 0

7. Secondary Outcome: Health Care Transition Feedback Survey: How Often do You Schedule Your Own Appointments With Your Health Care Provider?
Description: Specific item from the Health Care Transition Feedback Survey, created by Got Transition. The survey evaluated patients' experience with changing from a pediatric to an adult approach to care. This question evaluated how often the the patient scheduled their own appointments with their health care provider. Answer categories for this item were Always, Usually, Sometimes, and Never.
Time Frame: 12 months post-enrollment.
Population: Participants with survey data at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 51 | 26
Participants
  Always/Usually | 16 | 8
  Sometimes/Never | 35 | 18

8. Secondary Outcome: Health Care Transition Feedback Survey: Does Your Health Care Provider Update and Share a Medical Summary With You?
Description: Specific item from the Health Care Transition Feedback Survey, created by Got Transition. The survey evaluated patients' experience with changing from a pediatric to an adult approach to care. This question evaluated if the health care provider updated and shared a medical summary with the patient. Answer categories for this item were Yes or No.
Time Frame: 12 months post-enrollment.
Population: Participants with survey data at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 51 | 26
Participants
  Yes | 46 | 25
  No | 5 | 1

9. Secondary Outcome: Number of Ambulatory Visits Per Year
Description: Ambulatory visits was calculated for each patient as the average number of ambulatory visits per year. Ambulatory visits were identified by manual chart reviews and included primary care visits, visits with the hematology/SCD provider, and other outpatient specialty visits. Ambulatory visits per year was calculated as the total number of ambulatory visits reported over the duration of time on study (from enrollment to discontinuation of study participation).
Time Frame: Duration of time on study up, on average 23 months
Population: All enrolled subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: visits per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 196 | 95
visits per year | 5.31 [4.20 to 6.71] | 5.97 [4.62 to 7.71]

10. Secondary Outcome: Number of Visits With Adult Provider
Description: Adult provider visits was calculated for each patient as the average number of ambulatory visits that occurred with adult providers. These visits were identified by manual chart reviews. Adult provider visits per year was calculated as the total number of adult provider visits reported on study over the time from first visit with adult provider to end of study participation.
Time Frame: Adult duration of time on study, on average 16.5 months
Population: Among those with at least one visit with adult provider.
Measure: Least Squares Mean (95% Confidence Interval); unit: visits per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 147 | 32
visits per year | 6.16 [4.53 to 8.36] | 6.23 [4.27 to 9.10]

11. Secondary Outcome: Number of Hospitalization Days
Description: Hospitalization days was calculated for each patient as the average number of days spent inpatient for hospitalization per year. Inpatient dates were identified by manual chart reviews. Hospitalization days per year was calculated as the total number of hospitalization days reported on study over the total duration on study (from enrollment to discontinuation of study participation).
Time Frame: Duration of time on study, on average 23 months
Population: All enrolled subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: days per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 196 | 95
days per year | 4.38 [2.99 to 6.43] | 4.57 [3.05 to 6.84]

12. Secondary Outcome: Number of 14-day Readmissions
Description: 14-day readmissions was calculated for each patient as the number of hospital admissions that occur within 14 days after discharge from a previous admission, per year. Hospital admissions were identified by manual chart reviews and total number of readmissions within 14 days were counted over the duration of time on study.
Time Frame: Duration of time on study, on average 23 months.
Population: All enrolled subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: readmissions per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 196 | 95
readmissions per year | 0.14 [0.07 to 0.27] | 0.16 [0.07 to 0.33]

13. Secondary Outcome: Number of 30-day Readmissions
Description: 30-day readmissions will be calculated for each patient as the number of hospital admissions that occur within 30 days after discharge from a previous admission, per year. Hospital admissions were identified by manual chart reviews and total number of readmissions within 30 days were counted over the duration of time on study.
Time Frame: Duration of time on study, on average 23 months
Population: All enrolled subjects
Measure: Least Squares Mean (95% Confidence Interval); unit: readmissions per year
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
Number analyzed (Participants) | 196 | 95
readmissions per year | 0.25 [0.14 to 0.45] | 0.25 [0.13 to 0.49]

ADVERSE EVENTS:
Time Frame: All cause mortality was captured during the duration of time on study, an average of 23 months.
Description: Adverse event data were not collected due to the pragmatic nature of the trial, therefore the number of participants at risk for Serious Adverse Events and Other Adverse Events was zero. Deaths on study were captured and therefore All Cause Mortality is reported.
Arm/Group | Program Structured Education Based Transition Program | Structured Education Based Transition Program + Peer Mentoring
All-Cause Mortality (participants affected / at risk) | 2/196 | 3/95
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Because we did not complete enrollment and had imbalances in enrollment over time between the arms, we are not reporting p-values for comparisons between arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT03593395/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/95/NCT03593395/ICF_000.pdf